CLINICAL TRIAL: NCT03381768
Title: PD-L1 and PD-L2 Peptide Vaccination as Consolidation for Relapsed Follicular Lymphoma
Brief Title: Peptide Vaccination Against PD-L1 and PD-L2 in Relapsed Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lars Møller Pedersen (Other)
Responsible Party: Sponsor-Investigator, Lars Møller Pedersen, Chief consultant, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL1701; 2017-002000-28 (EudraCT Number)
Record Dates: First submitted 2017-12-08; First posted 2017-12-22 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Follicular Lymphoma
Keywords: PD-L1; PD-L2; peptide vaccine
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Programmed Cell Death 1 Ligand 2 Protein

STUDY DESIGN:
Intervention Model Description: Fixed dose safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): 3 vaccines of PD-L2 peptide followed by 12 vaccines of PD-L2 and PD-L1 peptide, over the course of one year.
  Interventions: Biological: PD-L2 peptide; Biological: PD-L2 and PD-L1 peptide

INTERVENTIONS:
Biological: PD-L2 peptide — 100 ug PD-L2 peptide dissolved in DMSO and water mixed with 500ul montanide.
Biological: PD-L2 and PD-L1 peptide — 100 ug PD-L2 peptide and 100ug PD-L1 peptide dissolved in DMSO and water mixed with 500ul montanide.

SUMMARY:
An open phase-1, first-in-human, clinical trial investigating the safety and immunological effects of peptide vaccination with Programmed Death Ligand 1 and 2 (PD-L1 and PD-L2) peptides in patients with relapsed follicular lymphoma.

DETAILED DESCRIPTION:
Follicular lymphoma (FL) is the the most common of the indolent lymphomas, with an incidence in Denmark of 220 per year. In 90% of the cases the disease is incurable why the treatment strategy often is watchful waiting until significant signs of progression or transformation. After chemotherapy, maintenance therapy is often used to increase disease control.

The microenvironment and immune escape mechanism are believed to play a major role in the persistence of the lymphoma. One escape mechanism is the PD-L1 and PD-L2 molecules expressed in the microenvironment of follicular lymphoma inhibiting the T-cells. By stimulating the T-cells to attack PD-L1 and PD-L2 expressing cells we hope to hamper the immunosuppressive tumor environment and establish immune tumor control.

10 patients treated with standard therapy are needed for the trial and each patient will receive 15 vaccinations over the course of one year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented FL grade I-IIIa, with no sign of current transformation. Patients cured of transformed lymphoma are eligible.
* A minimum of one line of induction therapy. Maintenance rituximab can continue along with the vaccination
* At least partial response to the latest standard treatment
* A minimum of 4 weeks since last treatment
* Age ≥ 18
* ECOG performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Progression with the presence of at least one GELF criteria or transformation at inklusion time.
* Other active malignant diseases
* Significant medical condition per investigators judgement e.g. severe Asthma/COLD, poorly regulated heart condition, insulin dependent diabetes mellitus.
* Acute or chronic viral/bacterial infection e.g. HIV, CMV, EBV, hepatitis or tuberculosis
* Serious known allergies or earlier anaphylactic reactions.
* Known sensibility towards Montanide ISA-51
* Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Adverse events evaluated by CTCAE 4.03 | 1 year follow up
  Adverse events are graded 1-5 according to the criteria

SECONDARY OUTCOMES:
Immune responses | 1 year
  T-cell cytokine release towards target antigens

OTHER OUTCOMES:
Clinical response according to Lugano criteria | 1 year
  Changes in tumor size on CT
Clinical response according to Lugano criteria | 1 year
  Changes in tumor metabolism on PET
Minimal residual disease | 1 year
  measured by circulating tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Klausen, MD, Principal Investigator — Hematological department, Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, RegionH, Denmark

IPD SHARING:
Plan to Share IPD: No